CLINICAL TRIAL: NCT00327067
Title: Iron Replacement in Blood Donors
Status: Completed | Type: Observational
Sponsor: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 060166; 06-CC-0166
Record Dates: First submitted 2006-05-17; First posted 2006-05-18 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-03-01

CONDITIONS: Iron Deficiency
Keywords: Hemoglobin; Iron Supplementation; Donor Retention; Iron Stores; Ferritin; Transferrin Saturation; Healthy Volunteer; HV; Blood Donors
MeSH Terms: conditions — Iron Deficiencies

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
Blood donors who have a low fingerstick hemoglobin level are usually deferred from donating. A possible solution to the problem of repeated deferrals might be for Blood Banks to offer donors with low hemoglobin levels oral iron supplements. To determine the feasibility of such a program, this study will:

* Determine the frequency of iron deficiency in first-time and repeat blood donors
* Examine the effects of long-term blood donation on donor hemoglobin levels and iron stores
* Compare body iron stores in donors who have low hemoglobin values with that of donors who have acceptable hemoglobin values at the time of donation
* Determine what conditions other than iron deficiency lead to low hemoglobin levels in blood donors
* Determine the safety and effectiveness of giving oral iron tablets to donors with low hemoglobin levels
* Monitor the effect of oral iron administration on donor satisfaction and donor retention.

First-time and repeat blood donors at the NIH Clinical Center Blood Bank 18 years of age and older may be eligible for this study. Participants include prospective donors who have an acceptable hemoglobin value at the time of donation and those whose hemoglobin level is determined to be too low for donation.

All participants do the following:

* Answer medical questions about their diet, health, and family history of blood disorders.
* Have blood samples drawn from their arm for testing blood cell counts, iron stores, and other hemoglobin-related tests as appropriate.

Donors with low hemoglobin also:

* Take iron supplements (ferrous sulfate) to replenish iron stores. (Donors who have previously had unpleasant side effects from ferrous sulfate are offered ferrous gluconate as an alternative.)
* Undergo evaluation with medical screening and laboratory tests at the time of future blood donations.

DETAILED DESCRIPTION:
Iron is an essential element that is lost with each blood donation. In order for a donor to compensate for the iron lost in donating blood, iron is mobilized from the body's iron stores and absorption of iron from the diet is increased. However, this balance is often difficult to maintain in premenopausal women and regular blood donors since there is ongoing blood loss. Deficiency in iron results in reduced hemoglobin values, iron stores, and eventually iron deficiency anemia if not treated. Iron deficiency presents a problem in blood centers since the minimum allowable hemoglobin for blood donation is 12.5 g per dL.

In the Department of Transfusion Medicine at the NIH, 14.6% of donors presenting for whole blood donation and 7.7% of donors presenting for apheresis platelet donation are deferred on at least one occasion per year due to low hemoglobin values. Overall, 7.9% of visits for whole blood donation and 2.1% of visits for apheresis platelet donation result in donor deferral due to low hemoglobin. Although the challenge of iron depletion in the blood donor population has been known for decades, little has been undertaken to resolve this issue. Several authors have reported data from successful short term projects demonstrating the safety and efficacy of iron replacement in donors, but larger long term studies have not been reported.

The objectives of this protocol are to: (1) quantitate the prevalence of iron deficiency in first-time presumably healthy individuals who present for blood donation; (2) study the effects of long-term blood donation on donors' hemoglobin levels and iron stores; (3) evaluate the safety, practicality, and efficacy of distributing oral replacement iron to blood donors; (4) determine the effect of oral iron replacement therapy on the donor pool by monitoring deferral rates for low hemoglobin before and after the initiation of an iron replacement program. The goal of these objectives is to treat and prevent iron deficiency in prospective and regular blood donors, thereby expanding the eligible donor pool and leading to increased donor satisfaction and retention by decreasing deferral rates due to low hemoglobin.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Subjects must meet all allogeneic donor eligibility criteria established by the NIH Department of Transfusion Medicine, American Association of Blood Banks, and the Food and Drug Administration
* Subjects must meet all research donor eligibility established by the NIH Department of Transfusion Medicine, per protocol 99-CC-0168
* Subjects must be 18 years of age or older
* Subjects must be willing to sign consent and participate in the protocol

EXCLUSION CRITERIA:

* Ineligible for volunteer or research blood donation, per DTM, AABB, or FDA criteria
* Subjects who refuse to sign the protocol consent document
* Subjects diagnosed with hereditary hemochromatosis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1820 (Actual)
Dates: Start 2006-05-12; Study Completion 2012-03-01

CONTACTS AND LOCATIONS:
Overall Officials: Stephen J O'Brien, Ph.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Davey RJ. Recruiting blood donors: challenges and opportunities. Transfusion. 2004 Apr;44(4):597-600. doi: 10.1111/j.0041-1132.2004.04402.x. No abstract available. PMID 15043578
- [Background] Gordeuk VR, Brittenham GM, Hughes MA, Keating LJ. Carbonyl iron for short-term supplementation in female blood donors. Transfusion. 1987 Jan-Feb;27(1):80-5. doi: 10.1046/j.1537-2995.1987.27187121482.x. PMID 3810831
- [Background] Radtke H, Tegtmeier J, Rocker L, Salama A, Kiesewetter H. Daily doses of 20 mg of elemental iron compensate for iron loss in regular blood donors: a randomized, double-blind, placebo-controlled study. Transfusion. 2004 Oct;44(10):1427-32. doi: 10.1111/j.1537-2995.2004.04074.x. PMID 15383014